CLINICAL TRIAL: NCT04810039
Title: Comparison of the Accuracy of the Neurological Prognosis at 6 Months of Traumatic Brain Injury Between Junior and Senior Doctors.
Acronym: PREDICT II
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210394
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-04

CONDITIONS: Prognosis of Neurological Outcome at 6 Months in Patients Undergoing Traumatic Brain Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- doctor working in neuro-intensive unite care: doctor predicting the outcome of the Glasgow Outcome Scale (GOS) score at 6 months compared to the actual outcome, in 20 anonymized records.
  Interventions: Other: Predict the outcome of the Glasgow Outcome Scale

INTERVENTIONS:
Other: Predict the outcome of the Glasgow Outcome Scale — Predict the outcome of the Glasgow Outcome Scale (GOS) score at 6 months compared to the actual outcome, in 20 anonymized records.

SUMMARY:
PREDICT II is an observational, prospective design, single-center study aiming to determine whether the prognosis of neurological outcome at 6 months in patients undergoing traumatic brain injury established by a doctor at his initial management is more accurate in experienced doctors versus junior doctors.

DETAILED DESCRIPTION:
Head injury is a non-rare cause of mortality and morbidity in young adults. It is difficult and often uncertain to assess the long-term neurological prognosis in these patients. However, this element is of major importance because it allows the clinician to determine the intensity of the therapies used and to adapt the information given to the patient and his relatives.

Numerous studies have been carried out to study the prognosis of these patients, of which two are the most important: CRASH-study and IMPACT-study. However, of all these studies, none of them had the objective of comparing whether the experience of the clinician influenced the accuracy of his prognosis. Similarly, the PREDICT-TBI study conducted at our center, which aimed to compare the clinician's assessment with a prognostic score already in use (IMPACT score) for determining the prognosis of the brain injured person, did not study the influence of the clinician's experience on the accuracy of the prognosis.

Assessment of clinicians' judgment of neurological outcome in 20 patient charts.

20 records will be randomly selected from the N patients included in the PREDICT-TBI study.

These 20 pseudonymities records will be presented, including admission scans and pre-hospital clinical data.

For each clinician included, a questionnaire of the assumed neurological outcome of each patient will be completed and compared with the true neurological outcome, the main variable being the GOSE neurological outcome at 6 months (already collected in the PREDICT-TBI study).

Our hypothesis is that clinicians have a reliable judgment of the neurological outcome of the patient by estimating the probability of error of 30% in senior physicians and 40% in junior physicians. The reliability of this judgment will be measured by assessing the number of errors each clinician will make on the 20 medical records.

The main issue of the study is to better understand the prognosis at the initial phase in order to adapt the nature of the information given to the families in terms of prognosis.

The number of subjects needed is calculated by simulating two-sided tests of a generalized binomial model that compares the "senior" group to the "junior" group on 10,000 samples made up of n * 2 binomial variables (n = 20, probability of error in seniors p1 = 0.3 (PREDCIT-TBI) and p2 = 0.4 for juniors). With an alpha risk of 5%, a power of 80%, we calculate the n = 18 physicians per group.

Inclusion and consent: After obtaining their consent we will include 18 doctors per group spread over several establishments.

Methodology: We will randomly select 20 files of moderate or severe traumatic brain injury patients treated in the neuro-ICU department of the Pitié-Salpêtrière hospital between March 2019 and December 2020 and included in the PREDICT-TBI study (CPP no. 19.01.21.68040) after having obtained their non-opposition from themselves or from their trusted person and not having been the subject of a limitation of active therapies during the first 24 hours. The patient was also not the victim of a lack of care during the first 24 hours. The prognostic data recognized in the literature for the first 24 hours of treatment are found in the computerized medical records of METAVISION and Carestream. This data, after being anonymized, will be submitted to the clinician for evaluation during an interview of a predefined duration. The prognosis will be assessed by means of a questionnaire submitted to all physicians detailed in the appendix. Then, it will be compared to the effective neurological status 6 months after the trauma assessed by a phone interview with the patient himself or his relatives.

ELIGIBILITY:
Inclusion Criteria:

* Senior group: intensive care anaesthesists with more than 4 years of experience in neuro-intensive care unit
* Junior group : advanced semester intensive care anaesthesists interns at the end of an internship composed of 5 months specialized in neuro-ICU

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The senior group will be made up of intensive care anaesthesists with more than 4 years of experience in neuro-intensive care unit, and the junior group, of advanced semester intensive care anaesthesists interns at the end of an internship composed of 5 months specialized in neuro-ICU.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the number of errors the doctor makes when predicting the outcome of the Glasgow Outcome Scale (GOS) score at 6 months compared to the actual outcome, in 20 anonymized records | Baseline (At inclusion of physicians) or minimum 6 month after patient inclusion
variability between physicians | Baseline (At inclusion)
  We will ask the intensivists for each patients' data the patient's risk of becoming GOS < 4 at 6 months between 0 and 100. This measure will be analyzed as a response variable (16*38 = 576 assessments) in a three-level hierarchical linear mixed model. We will introduce random intercepts for patients within the intensivists and we will add fixed effects as the patient's real becoming and the intensivist's seniority. This model will yield an estimate of a variance between intensivists and another method to test the effect of seniority to determine the patient's becoming. We will carry out analysis with nlme package in R.
confidence in their prognosis | Baseline (At inclusion)
  measured with the multiple choice question: "How confident are you in the prognosis you just made?" and possible answers: Certain, Very confident, Confident, Not Confident, Unsure.
the information offered to relatives | Baseline (At inclusion)
  measured with the multiple choice question: " The family arrives distressed ond would like more information on the prognosis and disability at 6 months. You are the first point of contact. Do you insist on?" and possible answers: "The good prognosis factors", "prognostic uncertainty", "disability or possible death".

CONTACTS AND LOCATIONS:
Locations (1):
- Réanimation neurochirurgicale, Hôpital Pitié-Salpêtrière, Paris, France